CLINICAL TRIAL: NCT00444431
Title: Ureteropelvic Junction Obstruction in Early Childhood: Comparison of Surgical Therapy and Surveillance in Children With Scintigraphically Prooved Obstruction. A Prospective, Randomized, Controlled Multi-Center Study
Brief Title: Ureteropelvic Junction Obstruction in Early Childhood: Comparison of Surgical Therapy and Surveillance. A Prospective, Randomized, Controlled Multi-Center Study
Acronym: TOKU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-004090-13
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2007-03-07 (Estimated); Status verified 2007-03

CONDITIONS: Unilateral Ureteropelvic Junction Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Pyeloplasty

SUMMARY:
In this randomized trial surgical therapy and surveillance of ureteropelvic junction obstruction will be compared, regarding partial renal function.

ELIGIBILITY:
Inclusion Criteria:

* unilateral ureteropelvic junction obstruction
* diameter of renal pelvis greater 12 mm
* partial renal function of 35%-55% proofed by scintigraphy
* urodynamically relevant decrease in renal drainage proofed by diuresis scintigraphy at the age of 4 weeks up to 6 months
* Abscence of clinical symptoms
* Healthy contralateral kidney

Exclusion Criteria:

* Global decrease in renal function
* renal dystopia
* megaureter
* vesico-ureteral reflux
* progressive hydronephrosis
* oligohydrammnion
* voiding dysfunction
* bilateral hydronephrosis
* severe chronical illness
* decrease of partial renal function of more then 5% during allocation

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240
Dates: Start 2007-03

PRIMARY OUTCOMES:
partial renal function

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Rübben, Prof., Principal Investigator — University Hospital, Essen; Peter Hoyer, Prof., Principal Investigator — University Hospital, Essen
Locations (2):
- Germany (2):
  - University Hospital of Essen, Department of Pediatric Nephrology, Essen, North Rhine-Westphalia
  - University Hospital of Essen, Department of Urology, Essen, North Rhine-Westphalia